CLINICAL TRIAL: NCT02490293
Title: Is it Fair to Use Antibiotics After Laparoscopic Cholecystectomy for the Patients With Acutely Inflamed Gallbladder?; a Multicenter Randomized Controlled Trial
Brief Title: Is it Fair to Use Antibiotics After Laparoscopic Cholecystectomy for the Patients With Acutely Inflamed Gallbladder?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taeho Hong (Other)
Collaborators: Incheon St.Mary's Hospital (Other); Bucheon St. Mary's Hospital (Other); Uijeongbu St. Mary Hospital (Other); Catholic University of Korea Saint Paul's Hospital (Other)
Responsible Party: Sponsor-Investigator, Taeho Hong, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Seoul-05
Record Dates: First submitted 2015-06-15; First posted 2015-07-03 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Acute Cholecystitis
MeSH Terms: conditions — Cholecystitis, Acute | interventions — Cephalosporins; Saline Solution; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (cephalosporin) (Experimental): During the period of hospitalization, intake of active drug ('pacetin', 2nd generation cephalosporin). 3 g per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 500mg each (1 pill of cefaclor, the 2nd generation cephalosporin every 12 hrs) for three days.
  Interventions: Drug: Cephalosporin
- Group B (placebo) (Placebo Comparator): During the period of hospitalization, Intake of placebo (normal saline). 30cc per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 1000mg each (2 pill of vitamin C every 12 hrs) for three days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cephalosporin — During the hospitalization, intake of pacetin, 2nd generation cephalosporin. 3 g per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 500mg each (1 pill of cefaclor, the 2nd generation cephalosporin every 12 hrs) for three days.
  Other Names: 'Pacetin'
  Arms: Group A (cephalosporin)
Drug: Placebo — During the period of hospitalization, Intake of placebo (normal saline). 30cc per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 1000mg each (2 pill of vitamin C every 12 hrs) for three days.
  Other Names: normal saline and vitamin C
  Arms: Group B (placebo)

SUMMARY:
During the laparoscopic cholecystectomy for acute cholecystitis, most surgeons routinely use the postoperative antibiotics after surgery. However, there is no consensus regarding the actual need of postoperative antibiotics in these cases and the use of postoperative antibiotics remains controversial.

Investigators will compare the surgical outcomes after laparoscopic cholecystectomy to the patients who has no evidence of systemic infection, according to the usage of postoperative antibiotics or not. The investigators expect that the routine use of postoperative antibiotics after laparoscopic cholecystectomy for acute cholecystitis gallbladder will have no effects on the postoperative morbidity.

DETAILED DESCRIPTION:
Primary outcome of this study is the confirmation of safety in the cases of acute cholecystitis without postoperative antibiotics usage after laparoscopic cholecystectomy. For this purpose, the investigators compare the surgical infectious outcomes including the wound infection or abdominal infections according to the usage of postoperative antibiotics after laparoscopic cholecystectomy.

Secondary outcome of this study is the confirmation of efficacy according to skip the use of postoperative antibiotics after laparoscopic cholecystectomy.

The investigators estimate the efficacy using the comparing the outcomes such as duration of hospitalization according to the use of postoperative antibiotics or not.

ELIGIBILITY:
Inclusion Criteria:

* grade I Tokyo guideline for acute cholecystitis
* grade II Tokyo guideline for acute cholecystitis without the evidence of gallbladder perforation

Exclusion Criteria:

* chronic cholecystitis
* gallbladder polyp or gallbladder cancer
* the patient who underwent reduced port surgery
* the patient who underwent common bile duct exploration during the operation
* the patient who underwent concurrent operation
* the patient who had past history of upper abdominal surgery
* the patient who had a immunodeficiency state
* the case which had a suspicion of delayed bile leakage
* the case which had a incomplete cystic duct ligation
* the patient who underwent open conversion surgery during the operation
* the patient who had a high risk of bleeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Taeho Hong, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's hospital, Seoul, Seocho-gu, Banopo-dong, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A (Cephalosporin): During the period of hospitalization, intake of active drug ('pacetin', 2nd generation cephalosporin). 3 g per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 500mg each (1 pill of cefaclor, the 2nd generation cephalosporin every 12 hrs) for three days.
  Cephalosporin: During the hospitalization, intake of pacetin, 2nd generation cephalosporin. 3 g per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 500mg each (1 pill of cefaclor, the 2nd generation cephalosporin every 12 hrs) for three days.
- Group B (Placebo): During the period of hospitalization, Intake of placebo (normal saline). 30cc per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 1000mg each (2 pill of vitamin C every 12 hrs) for three days.
  Placebo: During the period of hospitalization, Intake of placebo (normal saline). 30cc per day divided into 3 times via intravenous route until the day of discharge.
  After discharge, oral intakes of 1000mg each (2 pill of vitamin C every 12 hrs) for three days.
Period: Overall Study
Arm/Group | Group A (Cephalosporin) | Group B (Placebo)
Started | 96 | 102
Completed | 94 | 99
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Cephalosporin) | Group B (Placebo) | Total
Number analyzed (Participants) | 93 | 95 | 188
Age, Categorical [Count of Participants; unit: Participants] — "Count of Participants", is available as an option in the drop down menu to more accurately describe the Measure Type in some cases.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 83 | 85 | 168
    >=65 years | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (15.3) | 52.0 (15.0) | 52.0 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 49 | 93
  Male | 49 | 46 | 95
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 93 | 95 | 188

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Infectious Postoperative Complications
Description: Incidence of infectious postoperative complications in patients who underwent a laparoscopic cholecystectomy due to grade I Tokyo guidelines for acute cholecystitis or grade II Tokyo guidelines for acute cholecystitis except the evidence of gallbladder perforation, with antibiotics or placebo
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Group A (Cephalosporin) | Group B (Placebo)
Number analyzed (Participants) | 93 | 95
Participants | 8 | 7

2. Secondary Outcome: Duration of Hospitalization
Description: the duration between the operation day and the day of discharge
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 2 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A (Cephalosporin) | Group B (Placebo)
Number analyzed (Participants) | 93 | 95
days | 3.5 (1.1) | 3.2 (1.0)

ADVERSE EVENTS:
Arm/Group | Group A (Cephalosporin) | Group B (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/95
Other Adverse Events (participants affected / at risk) | 14/93 | 14/95
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Cephalosporin) (N=93) | Group B (Placebo) (N=95)
pancreatitis (Gastrointestinal disorders) | 0 | 3
diarrhea (Gastrointestinal disorders) | 3 | 1
CBD stone (Hepatobiliary disorders) | 3 | 3
wound infection (Infections and infestations) | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No